CLINICAL TRIAL: NCT05056597
Title: Incentive Processing and Learning in Anorexia Nervosa and Bulimia Nervosa
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Christina Wierenga, Professor, University of California, San Diego
Other Study IDs: 800775
Record Dates: First submitted 2021-09-09; First posted 2021-09-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- AN-R: Participants that meet Diagnostic And Statistical Manual Of Mental Disorders (DSM-V) criteria for Anorexia Nervosa restricting subtype.
- AN-BP: Participants that meet DSM-V criteria for Anorexia Nervosa binging/purging subtype
- BN: Participants that meet DSM-V criteria for Bulimia Nervosa.
- Healthy Controls: Participants that do not meet DSM-V criteria for any disorder.

SUMMARY:
The purpose of this study is to investigate areas of the brain responsible for 'liking', 'wanting', and learning in adults with eating disorders using brain imaging techniques, computer tasks, a test meal, and self-report questionnaires and interviews. The investigators will study changes in brain activity using a procedure called functional magnetic resonance imaging (fMRI). This study will include 252 women with an eating disorder (63 AN-restricting type (AN-R), 63 AN-binge eating/purging type (AN-BP), 63 bulimia nervosa (BN)) and 63 healthy controls (HC) aged 18-39.

Aim 1: To examine neural differences in 'liking' and 'wanting' in ED relative to HC.

Aim 2: To examine differences in instrumental learning for reward and punishment in ED relative to HC.

Aim 3: To examine how 'liking' and 'wanting' drive instrumental learning in ED and predict clinical symptoms at baseline and 1 year later.

Exploratory Aim: To explore the associations of dopamine function, as measured by neuromelanin MRI (NM-MRI), with ED diagnosis and brain response to 'liking', 'wanting', and learning.

ELIGIBILITY:
Inclusion Criteria:

Eating Disorder Group:

* Between the ages of 18 and 39 years old
* Meet DSM-V criteria for AN-R, AN-BP, or BN

Healthy Control Group:

* Between the ages of 18 and 39 years old
* Have maintained 85% to 120% ideal body weight since menarche

Exclusion Criteria:

All Groups:

* Psychotic illness/other mental illness requiring hospitalization
* Current dependence on drugs or alcohol defined by DSM IV criteria. Additionally, positive test results for drug use on the day of the scan, apart of marijuana, will result in cancelling or rescheduling the scan because acute use will impact MRI measures.
* Physical conditions (e.g. diabetes mellitus, pregnancy) known to influence eating or weight
* Neurological disorder, neurodevelopmental disorder, or history of head injury with >30 min loss of consciousness
* Any contraindication to undergoing an MRI
* Primary obsessive compulsive disorder or primary major depressive disorder

Additional Exclusion Criteria for ED Group:

-If taking other psychotropic medication, any change in dosage in the 2 weeks before scanning

Additional Exclusion Criteria for Healthy Control Group:

* Meet criteria for the diagnosis of any psychiatric disorder currently
* Any history of binge eating or purging behaviors, including self-induced vomiting, laxative or diuretic misuse
* Use of any psychoactive or other medication known to affect mood or concentration in the last 3 months

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will recruit 189 adult women currently ill with ED including anorexia nervosa, restricting type (AN-R, n=63), AN binge eating/purging type (AN-BP, n=63), and bulimia nervosa (BN, n=63) and 63 healthy control (HC) women between the ages of 18 and 39.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
BOLD response | 1 Year
  Brain activity associated with 'liking', 'wanting', and learning
Reward and Punishment Learning | 1 Year
  Task reinforcement learning rate in reward and punishment trials
Connectome-based predictive modeling (CPM) | 1 Year
  Functional connectivity maps from task-based fMRI data and clinical data

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Eating Disorders Treatment and Research Program, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided